CLINICAL TRIAL: NCT01946971
Title: Lansoprazole in Preterm Infants With Gastroesophageal Reflux
Brief Title: Lansoprazole in Preterm Infants With Gastroesophageal Reflux (GER)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Konect-LASP
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Premature Infants; Gastroesophageal Reflux
MeSH Terms: conditions — Premature Birth; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PL (Experimental): Placebo once a day orally for 7 days, then lansoprazole 1mg/kg once a day orally for 7 days
  Interventions: Drug: Lansoprazole; Drug: Placebo
- LP (Experimental): Lansoprazole 1mg/kg orally once a day for 7 days, then placebo orally once a day for 7 days
  Interventions: Drug: Lansoprazole; Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole
  Other Names: lanston LFDT
Drug: Placebo

SUMMARY:
This study is crossover study to evaluate safety and efficacy of lansoprazole in preterm infants with gastroesophageal reflux.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant
* symptoms suspecting gastroesophageal reflux

Exclusion Criteria:

* unstable general conditions due infection or acute illness
* congenital anomaly in upper gastrointestinal tract including esophagus
* drug history of H2, proton pump inhibitor, blocker during last 1 week
* medication of warfarin, carbamazepine, phenytoin, rifampin
* inappropriate clinical conditions judged by researchers

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Acid reflux time (%) | day 0, day 7, day 14
  measured by 24hr pH impedance monitor

SECONDARY OUTCOMES:
Acid reflux frequency | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
Composite score | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
Acid reflux fraction | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
acid bolus reflux time/%, | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
nonacid bolus reflux time/% | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
bolus reflux time/% | day 0, day 7, day 14
  measured by 24hr pH impedance monitor
I-GERQ GERD score | day 0, day 7, day 14
  I-GERQ GERD score chart (Infant Gastroesophageal Reflux Questionnaire Gastroesophageal Reflux Disease)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea